CLINICAL TRIAL: NCT06450730
Title: Effectiveness of a Combined mHealth Cognitive Behavioral Therapy Psychological Intervention to Improve Psychological Well-being in Young Patients With Type 1 Diabetes.
Brief Title: Effectiveness of a Combined mHealth-CBT Psychological Intervention to Improve Psychological Well-Being in Young Patients With T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Rosario Castillo-Mayén, Dr, Maimónides Biomedical Research Institute of Córdoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDI2019-107304RB-I00-BLS-T1D
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Cognitive-behavioral Therapy; mHealth interventions; Psychological well-being
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Psychological Well-Being | interventions — Amyloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT face-to-face + app (Experimental): Combines face-to-face CBT sessions with online activities and resources trough a mobile app
  Interventions: Behavioral: Cognitive-Behavioral Therapy: face-to-face + app
- TAU Group (No Intervention): TAU Group Patients of the control group continued their usual treatment.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy: face-to-face + app — This group will receive three 1-hour face-to-face CBT sessions (1,3,8). Participants will be involved in psychoeducation and practical activities related to psychological variables crucial for the adequate management of the disease (emotion regulation, self-efficacy, psychological flexibility, decision-making, etc.). These activities will include role-playing, discussions, and assignments to highlight the importance of emotions, thoughts, and healthy behaviors in managing diabetes and and their impact on the quality of life.
  For the online sessions, an app will be developed to complement the face-to-face intervention. Participants will engage in 5-weeks of exercises with weekly activities related to the intervention content (2,5,6,7). The structure of the activities will mirror that of the face-to-face sessions and will include tasks, self-report instruments, reinforcement and activity monitoring. In addition, the app will incoportate multiple resources (texts, slides, videos).
  Arms: CBT face-to-face + app

SUMMARY:
Type 1 diabetes (T1D) can lead to psychological adjustments that impact the acceptance and management of this health condition, as well as the overall quality of life of patients, especially among the young. Therefore, there is a need for psychological interventions aimed at enhancing the psychological well-being of children and adolescents with T1D. The goal of this non-randomized controlled trial is to evaluate whether a combined intervention comprising mHealth (using an app) and face-to-face psychological sessions based on Barlow's protocol and cognitive-behavioral therapy techniques (CBT) is effective in enhancing psychological well-being in children and adolescents with T1D. The main hypotheses are:

* H1: The primary results expected to be obtained are a significant increase in psychological well-being, which means a decreased diabetes distress (DDS) (H1a) an increased subjective well-being (PANAS) (H1b) and a better self-efficacy for managing their emotions (RESE) (H1c).
* H2: As secondary outcomes, it is also expected that the combined mHealth-CBT intervention would increase the level of positivity (P-Scale) (H2a), the self-esteem (RSES) (H2b) and the satisfaction with life (SWLS) (H2c).

ELIGIBILITY:
Inclusion Criteria:

* Girls and Boys with a diagnosis of T1D 6 - 18
* Having a smartphone compatible with the APP created used for the mHealth intervention and daily access to internet
* Having the required digital skills to follow the mHealth intervention
* Not currently participating in another clinical trial involving a psychological intervention

Exclusion Criteria:

* Girls and Boys with a diagnosis of T1D >18 years
* Not Having a smartphone compatible with the APP created used for the mHealth intervention and daily access to internet
* Currently participating in another clinical trial involving a psychological intervention

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Baseline, immediately after intervention and four months later (follow-up)
  Diabetes Distress Scale (DDS; Polonsky et al., 2005) is a Likert-type scale of 17 items that measures the level of emotional distress related to diabetes in individuals living with this chronic condition and how it impacts their quality of life. Scores ranges from 1 "not a problem" to 5 "very serious problem".
Regulatory Emotional Self-Efficacy | Baseline, immediately after intervention and four months later (follow-up)
  Regulatory Emotional Self-Efficacy scale (RESE; Caprara & Gervino, 2001).It is designed to assess an individual's perceived self-efficacy in managing negative and expressing positive emotions. It is a five-point scale (1 = not capable at all; 5 = completely capable) to 12 items distributed across two factors: positive affect expression (4 items) and negative affect expression, further divided into handling dejection and distress (4 items), and handling anger and irritation (4 items).
Positive Affect and Negative Affect | Baseline, immediately after intervention and four months later (follow-up)
  Positive Affect and Negative Affect Scale (PANAS; Watson et al., 1988) It is a Likert-type scale of 20-item (10 items for positive and 10 items for negative affect, that assesses the extent to which the participants experienced positive affect in the last 2 weeks. Rated on a 5-point scale from 1 "not at all" to 5 "very much". It has been validated in Spanish (López-Gomez, et al., 2015)

SECONDARY OUTCOMES:
Positivity | Baseline, immediately after intervention and four months later (follow-up)
  The Positivity Scale (P Scale; Zuffianò et al., 2019) evaluates the predisposition of people to estimate their life and their experiences from a positive perspective. It is an 8-item Likert-type scale, ranging from 1 "completely false" to 5 "completely true".
Self-esteem | Baseline, immediately after intervention and four months later (follow-up)
  Rosenberg self-esteem scale (RSES; Rosenberg, 1965). The RSES is a10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be uni-dimensional. All items are answered using a 4-point Likert scale format ranging from 1 "strongly disagree" to 5 "strongly agree".
Satisfaction with Life | Baseline, immediately after intervention and four months later (follow-up)
  Satisfaction with Life Scale (SWLS, Diener et al., 1985; Spanish adaptation by Atienza et al., 2000). The SWLS employs a 7-point Likert-style response scale with 5 items, ranging from 1 "completely disagree" to 5 "totally agree".

CONTACTS AND LOCATIONS:
Overall Officials: Bárbara Luque, PhD, Principal Investigator — Universidad de Córdoba; Carmen Tabernero, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Reina Sofía University Hospital, Córdoba, Spain